CLINICAL TRIAL: NCT02528695
Title: Adipose Tissue Imaging in Patients With Type 2 Diabetes, Pilot Study
Brief Title: Adipose Tissue Imaging in Type 2 Diabetes
Acronym: ATI-DM2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: NL44098.091.13
Record Dates: First submitted 2015-08-18; First posted 2015-08-19 (Estimated); Last update posted 2017-05-31 (Actual); Status verified 2016-04

CONDITIONS: Diabetes Mellitus Type 2
Keywords: 18F-FDG PET/CT; Adipose tissue; type 2 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Glucose Clamp Technique

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Healthy euglycemic clamp (Active Comparator): In 5 healthy volunteers an 18F-FDG PET/CT will be performed during an euglycemic clamp
  Interventions: Radiation: 18F-FDG PET/CT; Device: euglycemic clamp
- healthy hypoglycemic clamp (Active Comparator): In 5 healthy volunteers an 18F-FDG PET/CT will be performed during a hypoglycemic clamp
  Interventions: Radiation: 18F-FDG PET/CT; Device: hypoglycemic clamp
- Type 2 diabetes hypoglycemic clamp (Experimental): In 5 type 2 diabetes patients, an 18F-FDG PET/CT will be performed during a hypoglycemic clamp
  Interventions: Radiation: 18F-FDG PET/CT; Device: hypoglycemic clamp

INTERVENTIONS:
Radiation: 18F-FDG PET/CT — 18F-FDG PET/CT
Device: euglycemic clamp — euglycemic clamp
  Arms: Healthy euglycemic clamp
Device: hypoglycemic clamp — hypoglycemic clamp
  Arms: Type 2 diabetes hypoglycemic clamp; healthy hypoglycemic clamp

SUMMARY:
The metabolic function of different white adipose tissue depots in the body and its role in the development of type 2 diabetes (T2D) remains unclear. Several studies have used fluor-18 fluorodeoxyglucose positron emission tomography with computed tomography (FDG PET/CT) to image the metabolic activity of different adipose tissues in lean and obese healthy subjects and in patients with T2D with or without euglycaemic hyperinsulinemic clamping, describing differences in metabolic activity of visceral adipose tissue (VAT), subcutaneous adipose tissue (SAT) and gluteal-femoral adipose tissue (GFAT). Recently, FDG PET/CT showed high glucose uptake in VAT and SAT under unintentional hypoglycaemic conditions in a non-diabetic patient. Evaluation of potential differences in FDG uptake in white adipose tissue between healthy volunteers and T2D patients and between VAT, SAT and GFAT in these subjects under hyperinsulinemic hypoglycaemic conditions would be of great value in further exploring the pathogenesis of insulin resistance in T2D.

DETAILED DESCRIPTION:
Type 2 diabetes has become a worldwide epidemic with a prevalence of approximately 700,000 patients and an annual incidence of 70,000 in the Netherlands. The development of T2D depends on both genetic and nutritional factors and is characterized by insufficient insulin secretion by the pancreatic beta-cells and insulin resistance in liver, skeletal muscle and white adipose tissue. Insulin resistance often precedes beta-cell loss and is associated with central obesity, high blood pressure, hyperinsulinemia and dyslipidemia, all of which may lead to microvascular and cardiovascular complications.

White adipose tissue is increasingly considered a key metabolic organ in the development of insulin resistance. Especially the distribution of adipose tissue in the body is important. Indeed, visceral adipose tissue is a risk factor for coronary heart disease, certain cancers and T2D and associated with an increased cardiovascular and all-cause mortality, whereas excess of subcutaneous adipose tissue is not. There are distinct differences in the functional and hormonal characteristics of VAT and SAT, which may explain part of the mechanisms underlying the development of insulin resistance.

A more complete understanding of the molecular mechanisms that lead to T2D will enable the identification of individuals at highest risk, which could lead to more targeted prevention and pharmacological therapy.

FDG PET/CT is an established tomographic technique to image glucose metabolism with validated applications in oncology, infectious and inflammatory diseases, brain metabolism and cardiac viability. Several studies exploring the usefulness of FDG PET in imaging glucose metabolism in white adipose tissue reported lower overall glucose uptake in obese than in lean subjects. In both subject groups, glucose uptake was higher in VAT than in SAT. Glucose uptake in VAT and SAT was inversely related to insulin resistance, but uptake in GFAT was not. There are only few studies analyzing glucose uptake in patients with T2D with FDG PET/CT. In one study the impact of abdominal obesity and newly diagnosed T2D on insulin action in adipose tissue was evaluated, suggesting an excess of SAT to provide a sink for glucose, and thereby resulting in a compensatory decrease in insulin resistance. More research is needed to demonstrate the differences in glucose uptake in various adipose tissue depots in patients with T2D and correlate it with insulin resistance.

In order to keep glucose at a constant level during the FDG PET examination, usually a hyperinsulinemic euglycaemic glucose clamp is performed before scanning. Recently, a case-report was published describing an FDG PET/CT during an iatrogenic hypoglycemic state in a non-diabetic patient, which demonstrated remarkably increased glucose uptake in VAT and SAT. Based on this observation we hypothesize that glucose uptake during a hypoglycaemic state will be more pronounced in various adipose tissue depots. To our knowledge, this has not been performed in healthy volunteers or in patients with T2D. A controlled hypoglycemic state may be achieved by a hyperinsulinemic hypoglycaemic clamp, which has been used in several clinical studies. A demonstration of differences in FDG uptake in white adipose tissue between healthy volunteers and T2D patients and between VAT, SAT and GFAT under hypoglycaemic conditions would provide more insight in the glucose metabolism of adipose tissue and contribute to our understanding of insulin resistance in T2D. Even more importantly, this imaging technique might help to better characterise patients with T2D or patients at risk to develop T2D, and may thereby help to increase our understanding of the pathophysiology of T2D and the metabolic syndrome, which could lead to more targeted prevention in patients at risk and to personalised pharmacological therapy after the onset of clinically overt disease.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* BMI 27-40

For healthy volunteers:

* Fasting blood glucose < 6.1 mmol/L
* HbA1c < 42 mmol/mol (6%)

For T2D patients:

* Clinical overt Type 2 Diabetes
* on a glucose-lowering diet or on oral glucose-lowering medication
* T2D stable and under control for minimal 2 years
* HbA1c < 75 mmol/mol (9%)

Exclusion Criteria:

* Renal dysfunction
* Overt symptomatic neuropathy or proliferative retinopathy
* A history of cardiovascular disease complications (myocardial infarction, stroke, peripheral artery disease)
* Pregnancy or lactating
* Using subcutaneous insulin
* Incapability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2014-11; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Glucose uptake in adipose tissue measured by uptake of 18F-FDG on PET images | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Martin Gotthardt, Prof. Dr., Principal Investigator — Radboud University Medical Center
Locations (1):
- RadboudUMC, Nijmegen, Gelderland, Netherlands